CLINICAL TRIAL: NCT05491044
Title: A Study of Orelabrutinib in CLL/SLL Patients Who Are Slowly Responding to Ibrutinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Head of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Slowly responding switch IIT
Record Dates: First submitted 2022-08-01; First posted 2022-08-08 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: CLL/SLL
MeSH Terms: interventions — orelabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- orelabrutinib (Experimental): CLL/SLL patients who are slowly responding to ibrutinib are switched to orelabrutinib.
  Interventions: Drug: orelabrutinib

INTERVENTIONS:
Drug: orelabrutinib — Orelabrutinib 150mg po qd d1-28, up to 2 years or until disease progression, intolerable toxicity, death, informed consent withdrawal or lost of follow up (whichever occurs first).

SUMMARY:
This is a single arm, multi-center study to evaluate the efficacy and safety of orelabrutinib for Chronic lymphocytic lymphoma（CLL)/small lymphocytic lymphoma (SLL) patients who are slowly responding to Ibrutinib switched to Orelabrutinib.

DETAILED DESCRIPTION:
The eligible CLL/SLL patients who are slowly responding to Ibrutinib will be switched to Orelabrutinib treatment. The patients will receive Orelabrutinib 150mg oral daily (28 days/cycle) for up to 2 year or until disease progression, intolerable toxicity, death, informed consent withdrawal or lost of follow up (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old， male or female
* Diagnosed as CLL/SLL based on iwCLL2018 criteria
* Enhanced computed tomography/magnetic resonance imaging (CT/MRI) detection had measurable lesions: at least one lymph node had a maximum axis of more than 1.5 cm and had a measurable vertical dimension
* ECOG score 0-2
* Slowly responding to ibrutinib is defined as: patients only achieve SD after 3 cycles of ibrutinib treatment
* Life expectancy ≥6 months
* Adequate bone marrow reserve and adequate organ function
* Participant or his/her legal agent must be willing to sign a written informed consent document.

Exclusion Criteria:

* Evidence of active Richter's transformation or any evidence of disease progression on ibrutinib therapy.
* CNS involvement by CLL
* Present or prior history of other malignant neoplasms, unless radical treatment has been performed and there is no evidence of recurrence or metastasis in the last 5 years
* Uncontrolled or significant cardiovascular disease
* Active hemorrhage within 2 months prior screening
* Cerebral ischemic stroke or bleeding within 6 months prior screening
* Other surgery history within 6 weeks prior screening
* Uncontrolled active systemic fungal, bacterial, virus or other microbe infection, or intravenous injection of antibiotics needed
* Anti-tumor corticosteroids treatment 1 week prior orelabrutinib and anti-tumor herbal medicine treatment within 4 weeks prior screening
* Activated or uncontrolled hepatitis virus B infection (HBsAg positive with/or HBc Ab positive and HBV-DNA titration positive), HCV-RNA positive, HIV positive.
* Accepted live vaccine or immunization within 4 weeks prior screening
* Medium / strong inhibition or induction of cytochrome P450 CYP3A is needed.
* Allergy to orelabrutinib or the subsidiary (or supplementary) material (Hydroxypropyl methylcellulose acetate succinate, mannitol, cross-linked sodium carboxymethylcellulose, hydroxypropyl cellulose, silica and magnesium stearate)
* Obvious gastro-bowel disease which may influence the intaking, transportation or absorption of the drug, or total gastrectomy.
* Pregnant or breeding women, or women of childbearing age who are unwilling to take contraceptive measures during the whole study period and within 180 days after the last administration of the study drug; non surgically sterilized men who are unwilling to take contraceptive measures during the whole study period and within 180 days of the last administration of the study drug.
* Potentially life-threatening situation, or severe organ dysfunction, or situations the researchers think not suitable for the trial
* Any mental or cognitive impairment which may limit the understanding and implementation of informed consent or the compliance with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08-28 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
ORR at cycle 3 after switched to orelabrutinib | at cycle 3 (28 days/cycle)
  Overall response rate is defined as the proportion of patients with a best response of CR/CRi and PR/PR-L

SECONDARY OUTCOMES:
DOR | Up to 2 years
  The time from the first assessment of CR/CRi or PR/PR-L to progressive disease or death (due to any cause).
PFS | Up to 2 years
  Progression-free survival is calculated from the date of start of therapy until the date of first documented progress or death due to any cause.
OS | Up to 2 years
  Overall survival is defined as the duration from start of treatment to time of death.

OTHER OUTCOMES:
BTK occupancy | Before taking orelabrutinib and take orelabrutinib for 3-6 cycles
  The percentage of orelabrutinib/ibrutinib-bound BTK

CONTACTS AND LOCATIONS:
Overall Officials: Shenmiao Yang, Principal Investigator — Peking University People's Hospital
Locations (2):
- China (2):
  - Department of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No